CLINICAL TRIAL: NCT00842192
Title: A Prospective, Multicentre, Multinational, Open Label, Non-controlled, Observational, 24-week Study in Patients Using Oral Anti-Diabetic (OAD) Drugs + Levemir® (Insulin Detemir) for Treatment of Type 2 Diabetes Mellitus in Near East Region Countries
Brief Title: An Observational Study in Type 2 Diabetic Patients on Oral Antidiabetic Drugs and Basal Insulin in Near East Countries
Acronym: BO2NE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3735
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Insulin detemir for s.c. injection, once daily, in addition to current OAD treatment. Dose to be determined by physician.
  Other Names: NN304; Levemir®

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to investigate the safety and efficacy of insulin detemir as add-on therapy in type 2 diabetic patients who are using oral antidiabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* After the physician decision has been made to use insulin detemir therapy, any subject with Type 2 diabetes who is treated with any one or more of the oral antidiabetic drug (metformin, SU, repaglinide, TZDs) is eligible for the study. The selection of the subjects will be at the discretion of the individual physician. Particular attention should be paid to the drug interactions that are listed within the product label

Exclusion Criteria:

* Subjects currently being treated with insulin detemir or any other insulin regimen including regular(bolus) insulin
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 6 months. Women of childbearing potential who are not using adequate contraceptive methods

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 2 diabetes who is newly diagnosed or treated with OADs only is eligible for the study. The selection of the subjects as well as the treatment insulin will be at the discretion of the individual physician based on clinical judgement.
Sampling Method: Non-Probability Sample
Enrollment: 2155 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in number of hypoglycaemic events from baseline | at 12 and 24 weeks
HbA1c | at 12 and 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects to reach HbA1c between 6.5 and 7.0% | at 12 and 24 weeks
Glucose variability as measured by FPG | at 12 and 24 weeks
Postprandial glycaemic control as measured by PPG | at 12 and 24 weeks
Insulin dose and number of injections | at 12 and 24 weeks
Body weight | at 12 and 24 weeks
Number of adverse drug reactions (ADR) | at 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Amman, Jordan
- Novo Nordisk Investigational Site, Amman, Lebanon
- Novo Nordisk Investigational Site, Karachi, Pakistan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com